CLINICAL TRIAL: NCT01506466
Title: Weight Variation and Mechanisms Involved, During Chemotherapy in Breast Cancer Patients
Brief Title: Weight Variation During Chemotherapy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-A00206-35
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: chemotherapy; metabolism; weight; body composition
MeSH Terms: conditions — Breast Neoplasms; Body Weight | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- additional examinations/measurements (Other)
  Interventions: Other: blood test/ additional measurement

INTERVENTIONS:
Other: blood test/ additional measurement — blood test (hormonal, inflammatory, lipid and growth factors); body composition measurements; energy balance evaluation

SUMMARY:
Weight variation has been reported as a side effect of chemotherapy treatment in early breast cancer patients. To date, there is growing evidence for an increased risk of relapse and death in these patients who gain or lose weight. However, causes of weight variation during chemotherapy and mechanisms involved in the poor prognosis have been little studied.

Thus, the investigators are conducting a prospective study to characterize weight variation in terms of body composition and to identify the mechanisms involved.

ELIGIBILITY:
Inclusion Criteria:

* menopausal women
* breast cancer
* patients requiring chemotherapy treatment
* WHO performance status 0-2

Exclusion Criteria:

* diabetics
* patients with metastases
* other cancer

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body composition | within 2 weeks before chemotherapy; 1month after the last chemotherapy; and 6 months later.

SECONDARY OUTCOMES:
Change from baseline in energy balance | within 2 weeks before chemotherapy; 1month after the last chemotherapy; and 6 months later.
  resting energy expenditure, physical activity, food records.
Change from baseline in muscle strength | within 2 weeks before chemotherapy; 1month after the last chemotherapy; and 6 months later.
Change from baseline in biological factors (hormonal, inflammatory, lipid, growth factors) | within 2 weeks before chemotherapy; 1month after the last chemotherapy; and 6 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, MD, PhD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France